CLINICAL TRIAL: NCT00642733
Title: An Open Label Study to Evaluate the Effect of First Line Treatment With Tarceva in Combination With Gemcitabine on Overall Survival and Disease Progression in Patients With Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Brief Title: A Study of First Line Treatment With Tarceva (Erlotinib) in Combination With Gemcitabine in Patients With Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21285
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: gemcitabine

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 100mg po daily
Drug: gemcitabine — 1000mg/m2 iv weekly for 8 weeks, then weekly for 3 weeks of each 4 week cycle

SUMMARY:
This single arm study will assess the efficacy and safety of Tarceva + gemcitabine in patients with locally advanced, unresectable or metastatic pancreatic cancer. Patients will receive Tarceva 100mg po daily, in combination with gemcitabine 1000mg/m2 iv weekly for 8 weeks, followed by weekly for 3 weeks of each 4 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* pancreatic cancer, surgically unresectable or with metastases;
* no previous chemotherapy (except concomitant with radiotherapy);
* ECOG 0-2.

Exclusion Criteria:

* pancreatic cancer without histologic or cytologic confirmation;
* surgical resection possible;
* previous chemotherapy not concomitant with radiotherapy;
* ECOG 3-4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall survival; time to progression | 6 months

SECONDARY OUTCOMES:
Duration of response; disease-free survival | Event driven
AEs, lab parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Mexico (2):
  - Morelia
  - Tijuana